CLINICAL TRIAL: NCT04480905
Title: Effect of Dynamic Taping on Landing Kinematics and Kinetics in Volleyball Players With Symptoms of Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM109067F
Record Dates: First submitted 2020-07-01; First posted 2020-07-22 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Biomechanical Phenomena
Keywords: patellar tendinopathy; volleyball; biomechanics; kinematics; kinetics; dynamic tape; landing; VISA-P; translation; Chinese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tape group (Sham Comparator): in supine, full knee extension position, apply the sham tape from the anterior inferior iliac crest to the middle of the lower leg
  Interventions: Device: Sham tape
- Dynamic tape group (Experimental): in supine, full knee extension position, apply the dynamic tape from the anterior inferior iliac crest to the middle of the lower leg
  Interventions: Device: Dynamic tape

INTERVENTIONS:
Device: Dynamic tape — The dynamic tape will stick from anterior inferior iliac spine to the middle of the tibia in supine and full knee extension position
  Arms: Dynamic tape group
Device: Sham tape — The 3M™ Soft Cloth Tape will stick from anterior inferior iliac spine to the middle of the tibia in supine and full knee extension position
  Arms: Sham tape group

SUMMARY:
Patellar tendinopathy (PT) is the common cause of anterior knee pain, particularly in sports required repeated jumping and landing, such as volleyball. PT clinically presents as anterior knee pain and localized tenderness at the patellar tendon. To evaluate the severity of symptoms of PT, the VISA-P questionnaire is a self-administered, well-validated, and widespread assessment tool. In the long term, athletes would land with knee avoidance patterns and transfer the load to the hip joint caused further hip-related injury. Lower extremities eccentric exercise has been proven the most beneficial treatment of PT. However, the course lasts for three to six months. For athletes who are still in season, it's difficult to get the immediate effect. A newly developed biomechanical taping, dynamic tape, considered to be beneficial for load absorption during muscle eccentric contraction during landing and further normalized the lower extremities load contribution by its viscoelasticity property. However, no past research has confirmed this effect.

Therefore, the aims of the study are to translate the English VISA-P questionnaire to the Chinese and to study the reliability and validity of the Chinese version. In the next part, the investigators investigate the different landing biomechanics between individuals with and without patellar tendinopathy and establish the reliability of different landing tasks, and further explore whether the dynamic tape alters landing biomechanics in volleyball players.

DETAILED DESCRIPTION:
Patellar tendinopathy is one of the most common causes of anterior knee pain, particularly common in sports that required repeated jumping and landing, such as volleyball and basketball. Patellar tendinopathy clinically presents as anterior knee pain and localized tenderness at the patellar tendon. To evaluate the severity of symptoms of patellar tendinopathy, the VISA-P (Victorian institution of sports assessment- patellar tendon) questionnaire is an easily self-administered, well-validated assessment tool and commonly used across several countries. In the long term, athletes would land with knee avoidance landing patterns and transfer the load to the hip joint, which caused the further hip-related injury. Lower extremities eccentric contraction exercise has been proven the most beneficial treatment of patellar tendinopathy. However, the course of treatment needs to last for three to six months. For athletes who are still in season, it's difficult to get the immediate effect. A newly developed biomechanical taping, dynamic tape, considered to be beneficial for load absorption during muscle eccentric contraction during landing and further normalized the lower extremities load contribution by its viscoelasticity property. However, no past research has confirmed this effect.

Therefore, the aims of this study are to translate the English VISA-P questionnaire to Chinese and to study the reliability and validity of the Chinese version of the VISA-P. In the next part of the study, the investigators investigate the different landing biomechanics between individuals with and without patellar tendinopathy and establish the reliability of different landing tasks, and further explore whether the dynamic tape alters landing biomechanics in volleyball players. Methods: The first part of the study will include 15 subjects with the symptoms of patellar tendinopathy and 15 healthy subjects to fill out the translated questionnaire. In the second part of the study will include 15 volleyball players with the symptoms of patellar tendinopathy and 15 healthy controls. To compare the landing biomechanics between two groups, all subjects will conduct three landing tasks and the kinematics and kinetics of lower extremities、loading rate of vertical ground force and patellar tendon force will be recorded. In the third part of the study, the investigators will recruit 50 volleyball players with the symptoms of patellar tendinopathy and randomly assign to two groups, the dynamic tape, and sham tape. After taping, subjects will conduct three landing tasks, and the landing biomechanics will be recorded. Statistical analysis: Intra-class correlation, Pearson's correlation, and Mann-Whitney test will be used to analyze the test-retest reliability, concurrent validity, and construct validity of the Chinese version VISA-P. Repeated measures MANOVA will be used to analyze the interaction of landing biomechanics in three landing tasks between patellar tendinopathy group and healthy control, and further, analyze the interaction in three landing tasks between the dynamic tape and sham tape group in landing biomechanics parameters. Alpha level= 0.05

ELIGIBILITY:
Inclusion Criteria:

1. at the age of 16 to 35 years old
2. volleyball players joined the school team or professional level
3. over 90 minutes of training time per week -

Exclusion Criteria:

1. unbearable pain occurred at the patellar tendon when conducting landing tasks
2. there are currently other acute injuries to the lower extremity
3. lower extremity has undergone surgery or fracture in the past
4. with a history of rheumatoid arthritis, systematic and neurological diseases -

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
lower extremities joint angle | pre-intervention
  hip joint flexion, extension, abduction, adduction, internal rotation, external rotation angle, knee joint flexion, extension angle, ankle joint dorsiflexion, plantarflexion, inversion, eversion angle
lower extremities joint angle | immediately after the intervention
  hip joint flexion, extension, abduction, adduction, internal rotation, external rotation angle, knee joint flexion, extension angle, ankle joint dorsiflexion, plantarflexion, inversion, eversion angle
lower extremities joint angular velocity | pre-intervention
  hip joint flexion, extension, abduction, adduction, internal rotation, external rotation angle, knee joint flexion, extension angle, ankle joint dorsiflexion, plantarflexion, inversion, eversion angle divided by time
lower extremities joint angular velocity | immediately after the intervention
  hip joint flexion, extension, abduction, adduction, internal rotation, external rotation angle, knee joint flexion, extension angle, ankle joint dorsiflexion, plantarflexion, inversion, eversion angle divided by time
lower extremities joint angular acceleration | pre-intervention
  lower extremities joint angular velocity divided by time
lower extremities joint angular acceleration | immediately after the intervention
  lower extremities joint angular velocity divided by time
ground reaction force | pre-intervention
  anterior, posterior, medial, lateral, vertical ground reaction force
ground reaction force | immediately after the intervention
  anterior, posterior, medial, lateral, vertical ground reaction force
lower extremities joint force | pre-intervention
  calculate the reaction force between segments
lower extremities joint force | immediately after the intervention
  calculate the reaction force between segments
lower extremities joint moment | pre-intervention
  calculate the reaction moment between segments
lower extremities joint moment | immediately after the intervention
  calculate the reaction moment between segments
lower extremities joint power | pre-intervention
  calculate the reaction moment between segments
lower extremities joint power | immediately after the intervention
  calculate the reaction moment between segments
time to peak ground reaction force | pre-intervention
  time period from initial contact to peak vertical ground reaction force
time to peak ground reaction force | immediately after the intervention
  time period from initial contact to peak vertical ground reaction force
loading rate of ground reaction force | pre-intervention
  peak vertical ground reaction force divided by time to peak ground reaction force
loading rate of ground reaction force | immediately after the intervention
  peak vertical ground reaction force divided by time to peak ground reaction force
net joint work | pre-intervention
  integral of joint power over time
net joint work | immediately after the intervention
  integral of joint power over time
patellar tendon force | pre-intervention
  knee joint moment divided by moment arm
patellar tendon force | immediately after the intervention
  knee joint moment divided by moment arm

SECONDARY OUTCOMES:
lower extremities joint range of motion | before the landing tasks
  hip flexion, extension, internal rotation, external rotation, abduction, adduction, knee flexion, ankle plantar flexion, dorsiflexion, eversion, inversion joint range of motion measured by the physical therapist with a goniometer
lower extremities muscle force | before the landing tasks
  the hip flexor, extensor, internal rotator, external rotator, abductor, adductor, knee extensor, flexor, ankle plantar flexor, dorsiflexor, evertor, invertor muscle force measured by the physical therapist with a hand-held dynamometer
lower extremities muscle length | before the landing tasks
  iliopsoas, rectus femoris, hamstring, gastrocnemius and soleus muscle length test measured by the physical therapist

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, PhD, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No